CLINICAL TRIAL: NCT00476190
Title: ALL Adult Consortium Trial: Adult ALL Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Boston Children's Hospital (Other); NCIC Clinical Trials Group (Network)
Responsible Party: Principal Investigator, Daniel J. DeAngelo, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 06-254
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Doxorubicin; Cytarabine; Methotrexate; Vincristine; Cyclophosphamide; Hydrocortisone; Dexamethasone; pegaspargase; Imatinib Mesylate; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-amendment cohort, 2500 IU/m2 q2 weeks (Experimental): The first 66 patients enrolled under the initial design. In the post-induction phases, IV asparaginase was administered every two weeks at the higher dose of 2500 IU/m2, for a total of 30 post-induction weeks. IV asparaginase was administered as a single dose during induction. Protocol therapy was comprised of 6 phases: Prophase, Induction, Consolidation I, CNS, Consolidation II, and Continuation, and varied based off risk classification.
  Interventions: Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Methylprednisone; Drug: Hydrocortisone Sodium Succinate; Drug: Dexamethasone; Drug: 6-MP; Drug: PEG-Asparaginase; Drug: Imatinib; Drug: Etoposide; Procedure: Radiation Therapy; Drug: E. coli Asparaginase
- Post-amendment cohort, 2000 IU/m2 q3 weeks (Experimental): The 46 patients enrolled under amended design, after August 1, 2011. In the post-induction phases, IV asparaginase was administered every 3 weeks at the dose of 2000 IU/m2, for a total of 30 post-induction weeks. E. coli asparaginase was administered as a single dose during induction. Protocol therapy was comprised of 6 phases: Prophase, Induction, Consolidation I, CNS, Consolidation II, and Continuation, and varied based off risk classification.
  Interventions: Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Methylprednisone; Drug: Hydrocortisone Sodium Succinate; Drug: Dexamethasone; Drug: 6-MP; Drug: PEG-Asparaginase; Drug: Imatinib; Drug: Etoposide; Procedure: Radiation Therapy; Drug: E. coli Asparaginase

INTERVENTIONS:
Drug: Doxorubicin — Induction: Intravenously on days 4 and 5. Consolidation 1A: Intravenously on day 1. CNS Therapy: Intravenously on day 1. Consolidation II: Intravenously day 1 of each cycle.
Drug: Cytarabine — Prophase: Intravenously on days 1-3. Induction: Intrathecal on days 15 or 18. Consolidation IB: Intravenously or subcutaneous on days 2-5 and 9-12. Consolidation IC: Intravenously every 12 hours starting on day 1 CNS Therapy: Intrathecal 4 times over 2 weeks. Consolidation II: Intrathecal once every 18 weeks Continuation: Intrathecal every 18 weeks
Drug: Methotrexate — Induction: Intravenously on day 6 and intrathecally on day 29 or 32. Consolidation IA: Intravenously on day 1 and intrathecally on Day 1 (prior to IV).
  Consolidation IB: Intrathecally on day 1. CNS Therapy: Intrathecally 4 times over 2 weeks. Consolidation: Intrathecally once every 18 weeks. Continuation: Intravenously weekly and intrathecally every 18 weeks.
Drug: Vincristine — Induction: Intravenously on days 4, 11, 18, 25. Consolidation IA: Intravenously on day 1. CNS Therapy: Intravenously on day 1. Consolidation II: Intravenously on day 1 of each cycle.
Drug: Cyclophosphamide — Consolidation IB: Intravenously on day 1
Drug: Methylprednisone — Prophase: Intravenously on days 1-3
Drug: Hydrocortisone Sodium Succinate — Induction: Intrathecally on day 15 or 18. CNS Therapy: Intrathecally 4 times over 2 weeks. Consolidation II: Intrathecally once every 18 weeks. Continuation: Intrathecally every 18 weeks.
Drug: Dexamethasone — Consolidation IC: Orally on days 1-5 twice per day. Consolidation II: Orally on days 1-5 of each cycle. Continuation: Orally on days 1-5 of each cycle.
Drug: 6-MP — Induction: Orally on days 3-43 or 33-46. Consolidation IA: orally on days 1-14. Consolidation IB: orally on days 1-14. CNS Therapy: Orally on days 1-14. Consolidation II: Orally on days 1-14. Continuation: Orally on days 1-14 of each cycle.
Drug: PEG-Asparaginase — Consolidation IC: Intravenously every 3 weeks, starting on day 8. CNS Therapy: Intravenously every 3 weeks, starting 3 weeks after the Consolidation IC dose.
  Consolidation II: Intravenously every 3 weeks.
Drug: Imatinib — Used for PH+ ALL subjects enrolled prior to May 1st 2011 only and is used continuously throughout every phase of treatment.
Drug: Etoposide — Consolidation IC: intravenously on days 3, 4 and 5 of this cycle.
Procedure: Radiation Therapy — Given during CNS Therapy either 8 or 10 daily treatments, on days 1-8 or 1-10, depending upon leukemia involvement in the CSF
Drug: E. coli Asparaginase — Intramuscularly Day 7 of Induction.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a multi-drug chemotherapy regimen in adult patients with Acute Lymphoblastic Leukemia (ALL). We will use a regimen that is often used in pediatric patients and we will add drugs called PEG-asparaginase and E. coli asparaginase. PEG-asparaginase has been given as an injection in the past and has been used in treatment with both children and adults with ALL. Information from those other research studies suggests that intravenous PEG-asparaginase has been administered safely in both children and adults. We hope to gain more information about the participants disease and how it responds to standard chemotherapy drugs used to treat ALL>

DETAILED DESCRIPTION:
* This study has several periods of treatment called phases and uses several different drugs in each phase. The drugs may be given by mouth, into a vein, or into the spinal fluid (called intrathecal chemotherapy). In some individuals this treatment helps prevent leukemia cells from coming back in the spinal fluid and brain. Radiation therapy will also be administered as part of this treatment regimen.
* The treatment program consists of 2-different treatment arms with six separate phases of therapy. The phases of treatment are: (1) Steroid prophase (2) Induction (3) Consolidation I (4) Central nervous system (CNS) therapy (5) Consolidation II (6) Continuation.
* The participants treatment arm will depend on the status of their leukemia at the end of the induction therapy (the second phase of treatment). Arm A: all participants who achieve complete remission after Induction and Arm B: all participants who fail to achieve a complete remission after Induction.
* Steroid Prophase: All participants are involved in this treatment phase which consists of two drugs, one given intravenously (IV) and one given intrathecally. This phase lasts 3 days and the purpose is to collect scientific data that might be useful in the future and to see how steroids work in treating leukemia
* Induction: This phase begins immediately after the steroid prophase and lasts about 1 month. Induction is used to cause a remission. Eight drugs are used during this phase of treatment, and administration is either orally, IV or intrathecal. On day 29, participant's bone marrow and peripheral blood counts will be tested. If they have achieved complete remission or partial remission, they will proceed to the next phase of treatment. If they are not in complete remission, they will receive vincristine by IV on days 32, 39 and 46, until complete remission is achieved. If they do not achieve complete or partial remission by day 53 they will be removed from the study.
* Consolidation I: This phase of treatment begins as soon as there is a documented confirmation that the participant's leukemia is either in complete or partial remission. Treatment in this phase lasts about 7 weeks and is intended to further reduce the number of leukemia cells in the body. This consolidation treatment consists of 3 phases: 1A, 1B and 1C. Each phase involves a three week cycle of chemotherapy. Arm A and Arm B will be assigned according to remission status after induction therapy and will determine the order that the participant follows the Consolidation phases.
* Central Nervous System (CNS) Therapy: CNS therapy begins 3 weeks after the end of Consolidation I therapy and should last 3 weeks. Treatment includes a series of lumbar punctures with the administration of anti-leukemia drug as well as oral drugs and IV drugs. Radiation therapy will also be given during this phase of therapy. The purpose of radiation therapy is to prevent leukemia from coming back in the brain. Radiation therapy will be given in either 8 or 10 daily treatments.
* Consolidation II Therapy: This phase begins as soon as CNS therapy ends and lasts about 27-30 weeks. It consists of cycles of chemotherapy repeated every three weeks along with IV PEG-asparaginase administered every 3 weeks. The cycles will be repeated until the participant receives a total of 10 doses of asparaginase.
* Continuation Therapy: This phase begins after the end of the Consolidation II phase. The goal of this phase is to get rid of all leukemia in the body. It consists of cycles of chemotherapy repeated every three weeks and will last until the participant has been in remission for two years.
* During all phases of treatment, participants will have tests and procedures to monitor their health and for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia, excluding known mature B-cell ALL by the presence of any of the following: surface immunoglobulin, L3 morphology, t(8;14)(q24;q32), t(8;22), or t(2;8)
* Age 18.00-50.99 years

Exclusion Criteria:

* Prior anti-leukemic therapy except 1 week or less of steroids, and/or emergent radiation therapy to the mediastinum, or hydroxyurea or emergent leukopheresis
* Known HIV positive
* Secondary ALL
* Pregnant or breast feeding women
* Patients with an active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2007-04; Primary Completion 2013-09 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel DeAngelo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (15):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital of Boston, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - LDS Hospital, Salt Lake City, Utah
- Canada (8):
  - Vancouver Cancer Center, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII, Health Sciences Centre, Halifax, Nova Scotia
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Started | 66 | 46
Eligible and Treated | 65 | 45
Treated and Toxicity Data Reported | 66 | 44
Eligible and Treated and Toxicity Data Reported | 65 | 44
Evaluable for Complete Remission | 64 | 39
Achieved Complete Remission | 57 | 34
Proceeded to Stem Cell Transplant (SCT) | 15 | 6
Initiated Asparaginase Consolidation Therapy | 42 | 28
Completed | 25 | 20
Not Completed | 41 | 26
Not completed — Ineligible | 1 | 1
Not completed — Induction Death | 2 | 0
Not completed — Induction Failure | 2 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Relapse/Progression | 5 | 2
Not completed — Remission Death | 0 | 1
Not completed — Transplant in first Complete Remission (CR) | 15 | 6
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Other | 9 | 10

BASELINE CHARACTERISTICS:
Population: This analysis dataset is comprised of all eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks | Total
Number analyzed (Participants) | 65 | 45 | 110
Age, Customized [Count of Participants; unit: Participants]
  18-19 years | 6 | 3 | 9
  20-29 years | 20 | 18 | 38
  30-39 years | 19 | 11 | 30
  40-50 years | 20 | 13 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 40 | 27 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 56 | 37 | 93
  Unknown or Not Reported | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 58 | 30 | 88
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 5 | 10 | 15
Immunophenotype [Count of Participants; unit: Participants]
  B-cell | 56 | 34 | 90
  T-cell | 9 | 11 | 20
White Blood Count (WBC) (x10 ^-3) at diagnosis (cells/uL) [Count of Participants; unit: Participants]
  <30 | 48 | 33 | 81
  >=30 | 17 | 11 | 28
  Unknown | 0 | 1 | 1
Central Nervous System (CNS) status at diagnosis [Count of Participants; unit: Participants]
  CNS 1 (-) CSF WBC <5 without blasts | 40 | 37 | 77
  CNS 2 (+) CSF WBC <5 with blasts | 4 | 3 | 7
  CNS 3 (+) CSF WBC ≥5 with blasts | 2 | 2 | 4
  Traumatic Tap with Blasts | 5 | 0 | 5
  Traumatic Tap without Blasts | 12 | 2 | 14
  Not performed | 2 | 1 | 3
Eastern Cooperative Oncology Group (ECOG) Risk Classification [Count of Participants; unit: Participants] — ECOG risk is defined as follows: HR includes any patients with an MLL rearrangement or Ph+ and B-cell patients with WBC ≥ 35K or age ≥ 35 years and T-cell patients with WBC ≥ 100K.
  Participants
    Standard Risk (SR) | 31 | 25 | 56
    High Risk (HR) | 34 | 20 | 54

OUTCOME MEASURES:

1. Primary Outcome: Asparaginase Completion Rate
Description: Feasibility based on the rate of asparaginase completed defined as the percentage of patients who, after having achieved a complete remission after induction therapy, complete >25 weeks of IV PEG asparaginase as part of intensification therapy. Complete remission is defined as an interpretable bone marrow (a specimen with normal marrow elements present) with fewer than 5% lymphoblasts and peripheral blood without lymphoblasts, and an antigen presenting cell (APC) > 1000/mm3 and platelets > 100,000/mm3, and no evidence of extramedullary leukemia.
Time Frame: Assessed at the end of the 30-week post-induction treatment period or when the participant comes off treatment, whichever occurs first.
Population: The analysis dataset is comprised of all patients who initiated asparaginase consolidation therapy.
Measure: Number (80% Confidence Interval); unit: Percentage of patients
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Number analyzed (Participants) | 42 | 28
Percentage of patients | 43 [32 to 54] | 79 [65 to 88]

2. Primary Outcome: Number of Participants With Grade 3 or Worse Toxicity.
Description: Defined as the number of participants who experience the following grade 3 or worse adverse events based on Common Terminology Criteria for Adverse Events (CTCAE) v3: Neutrophils, Platelets, Febrile neutropenia, Infection, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Bilirubin, Liver dysfunction/failure, Hyperglycemia, Stomatitis, CNS hemorrhage, Thrombosis, Seizure, Osteonecrosis, Hypersensitivity, Pancreatitis, Neuropathy.
Time Frame: Assessed on an ongoing basis (at least once every 3 months) while on study, including the treatment phases of Induction, Consolidation I & II, CNS, and Continuation. Treatment duration for this study was a median (range) of 287 days (2-974).
Population: The analysis dataset is comprised of all eligible and treated patients for whom toxicity data is reported.
Measure: Number; unit: participants
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Number analyzed (Participants) | 65 | 44
participants
  Neutrophils | 49 | 31
  Platelets | 44 | 30
  Febrile neutropenia | 30 | 23
  Infection with grade 3/4 neutropenia | 24 | 10
  Infection, other | 5 | 3
  AST | 19 | 5
  ALT | 34 | 13
  Bilirubin | 24 | 3
  Liver dysfunction/failure | 2 | 1
  Hyperglycemia | 10 | 8
  Stomatitis | 8 | 2
  CNS hemorrhage | 2 | 0
  Thrombosis | 19 | 7
  Seizure | 5 | 0
  Osteonecrosis | 4 | 1
  Hypersensitivity | 3 | 6
  Pancreatitis | 1 | 2
  Neuropathy | 5 | 4

3. Secondary Outcome: Complete Remission Rate
Description: Complete remission rate is defined as the percentage of patients with an interpretable bone marrow (a specimen with normal marrow elements present) with fewer than 5% lymphoblasts and peripheral blood without lymphoblasts, and an antigen presenting cell (APC) > 1000/mm3 and platelets > 100,000/mm3, and no evidence of extramedullary leukemia.
Time Frame: 3-day Steroid prophase and 4-week induction treatment period. Participants are assessed on Day 32 of induction.
Population: The analysis dataset is comprised of all patients who are evaluable for complete remission
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Number analyzed (Participants) | 64 | 39
Participants | 57 | 34

4. Secondary Outcome: 3-year Disease Free Survival
Description: Disease-Free Survival (DFS) based on the Kaplan-Meier method is defined as the time from achieving a complete remission to the first of disease recurrence or death, censored at time of last disease assessment. 3-year DFS is the percentage probability of patients remaining alive, relapse-free and without occurrence of second malignant neoplasm 3 years from complete remission. Disease release is defined as >25% lymphoblasts identified morphologically in bone marrow aspirate/biopsy, or identification of lymphoblasts in marrow (any percentage) identified to be leukemic by flow cytometry, cytogenetics, fluorescent in situ hybridization (FISH), immunohistochemistry, or other tests. Appearance of leukemic cells at any extramedullary site (a single, unequivocal lymphoblast in the cerebrospinal fluid (CSF) may qualify as CNS leukemia) also qualifies if confirmed by the PI.
Time Frame: Assessed continuously throughout the treatment period, and annually for 5 years following the completion of protocol treatment (up to 5 years). Relevant for this measure is 3 years from the date of complete remission.
Population: The analysis dataset is comprised of all eligible patients who achieved a complete remission.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Number analyzed (Participants) | 57 | 34
Percentage of patients | 70 [56 to 81] | 75 [53 to 88]

5. Secondary Outcome: 3-year Overall Survival
Description: Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from study entry to death from any cause and will be censored the date last known alive.
Time Frame: Assessed continuously throughout the treatment period, and annually for 5 years following the completion of protocol treatment (up to 5 years). Relevant for this measure is 3 years from the date of study entry.
Population: The analysis dataset is comprised of all eligible patients.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
Number analyzed (Participants) | 65 | 45
Percentage of patients | 70 [57 to 80] | 83 [67 to 91]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were continuously monitored and reported every 3 months during treatment. Adverse events were monitored for the treatment duration of this study, which was a median (range) of 287 days (2-974). All-Cause Mortality was monitored for the duration of follow-up for this study, which was a median (range) of 3.27 years (0.01-11.8). Data is reported for the entire study cohort (n=112) and broken down by arm.
Description: Reporting included all observed adverse events, with grade and attribution to study treatment. Maximum grade by type was calculated with serious adverse events defined as either 1) G5, 2) G4 unless myelosuppression or unequivocally due to disease or considered expected for chemotherapy drugs used, 3) G2 or G3 events that are unexpected and Possibly, Probably, or Definitely related to study treatment. Since SAE data was not collected separately, all AEs have been reported in the SAE table.
Arm/Group | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks | Post-amendment Cohort, 2000 IU/m2 q3 Weeks
All-Cause Mortality (participants affected / at risk) | 24/66 | 12/44
Serious Adverse Events (participants affected / at risk) | 66/66 | 44/44
Other Adverse Events (participants affected / at risk) | 0/66 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-amendment Cohort, 2500 IU/m2 q2 Weeks (N=66) | Post-amendment Cohort, 2000 IU/m2 q3 Weeks (N=44)
Anemia (Blood and lymphatic system disorders) | 42 | 19
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 8 | 9
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 33 | 27
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 5 | 5
Chest pain - cardiac (Cardiac disorders) | 1 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 8 | 5
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 16 | 7
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 6 | 5
Ear pain (Ear and labyrinth disorders) | 3 | 3
External ear pain (Ear and labyrinth disorders) | 2 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 2
Adrenal insufficiency (Endocrine disorders) | 2 | 2
Cushingoid (Endocrine disorders) | 11 | 4
Endocrine disorders - Other, specify (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 7 | 6
Cataract (Eye disorders) | 1 | 2
Dry eye (Eye disorders) | 2 | 3
Extraocular muscle paresis (Eye disorders) | 3 | 2
Eye disorders - Other, specify (Eye disorders) | 12 | 6
Eye pain (Eye disorders) | 4 | 3
Flashing lights (Eye disorders) | 0 | 2
Papilledema (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 4 | 1
Watering eyes (Eye disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 8 | 4
Abdominal pain (Gastrointestinal disorders) | 40 | 24
Anal fistula (Gastrointestinal disorders) | 2 | 1
Anal pain (Gastrointestinal disorders) | 6 | 5
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 3
Colonic perforation (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 32 | 23
Dental caries (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 40 | 22
Dry mouth (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 25 | 14
Dysphagia (Gastrointestinal disorders) | 4 | 4
Enterocolitis (Gastrointestinal disorders) | 2 | 2
Esophageal pain (Gastrointestinal disorders) | 2 | 1
Esophageal ulcer (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 6 | 1
Fecal incontinence (Gastrointestinal disorders) | 5 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 20 | 17
Gingival pain (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 6 | 11
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 28 | 18
Nausea (Gastrointestinal disorders) | 55 | 37
Oral hemorrhage (Gastrointestinal disorders) | 3 | 0
Oral pain (Gastrointestinal disorders) | 6 | 9
Pancreatitis (Gastrointestinal disorders) | 4 | 3
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal pain (Gastrointestinal disorders) | 6 | 6
Stomach pain (Gastrointestinal disorders) | 1 | 4
Toothache (Gastrointestinal disorders) | 3 | 3
Typhlitis (Gastrointestinal disorders) | 3 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 48 | 24
Chills (General disorders) | 17 | 9
Death NOS (General disorders) | 2 | 0
Edema face (General disorders) | 3 | 2
Edema limbs (General disorders) | 34 | 14
Edema trunk (General disorders) | 5 | 1
Fatigue (General disorders) | 54 | 32
Fever (General disorders) | 19 | 16
Flu like symptoms (General disorders) | 3 | 2
Gait disturbance (General disorders) | 2 | 1
General disorders and administration site conditions - Other, specify (General disorders) | 12 | 12
Injection site reaction (General disorders) | 6 | 0
Localized edema (General disorders) | 4 | 0
Non-cardiac chest pain (General disorders) | 10 | 6
Pain (General disorders) | 27 | 15
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 4 | 1
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 5 | 1
Allergic reaction (Immune system disorders) | 12 | 15
Immune system disorders - Other, specify (Immune system disorders) | 2 | 2
Abdominal infection (Infections and infestations) | 1 | 0
Bone infection (Infections and infestations) | 1 | 0
Bronchial infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 5 | 0
Conjunctivitis infective (Infections and infestations) | 2 | 0
Encephalomyelitis infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 8 | 5
Eye infection (Infections and infestations) | 1 | 1
Gum infection (Infections and infestations) | 3 | 2
Infections and infestations - Other, specify (Infections and infestations) | 42 | 27
Kidney infection (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 5 | 2
Nail infection (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 1
Penile infection (Infections and infestations) | 1 | 0
Peripheral nerve infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 6 | 1
Sinusitis (Infections and infestations) | 3 | 6
Skin infection (Infections and infestations) | 6 | 3
Upper respiratory infection (Infections and infestations) | 9 | 9
Urinary tract infection (Infections and infestations) | 3 | 3
Vaginal infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 13 | 7
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 0
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 4 | 9
Intraoperative skin injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 6 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 2
Activated partial thromboplastin time prolonged (Investigations) | 7 | 0
Alanine aminotransferase increased (Investigations) | 45 | 23
Alkaline phosphatase increased (Investigations) | 14 | 5
Aspartate aminotransferase increased (Investigations) | 36 | 17
Blood bilirubin increased (Investigations) | 38 | 4
CPK increased (Investigations) | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 1
Cholesterol high (Investigations) | 12 | 5
Creatinine increased (Investigations) | 7 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1
Fibrinogen decreased (Investigations) | 20 | 12
GGT increased (Investigations) | 10 | 4
INR increased (Investigations) | 6 | 1
Investigations - Other, specify (Investigations) | 22 | 7
Lipase increased (Investigations) | 8 | 4
Lymphocyte count decreased (Investigations) | 14 | 14
Neutrophil count decreased (Investigations) | 49 | 31
Platelet count decreased (Investigations) | 47 | 32
Serum amylase increased (Investigations) | 4 | 3
Weight gain (Investigations) | 6 | 0
Weight loss (Investigations) | 14 | 4
White blood cell decreased (Investigations) | 20 | 17
Acidosis (Metabolism and nutrition disorders) | 5 | 1
Anorexia (Metabolism and nutrition disorders) | 34 | 15
Dehydration (Metabolism and nutrition disorders) | 6 | 6
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 33 | 15
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 3 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 23 | 16
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 16 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 2
Hypokalemia (Metabolism and nutrition disorders) | 23 | 12
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 4
Hyponatremia (Metabolism and nutrition disorders) | 14 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 8 | 4
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 3 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 22
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 18 | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 24 | 7
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 13 | 4
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 20 | 8
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 12
Neck pain (Musculoskeletal and connective tissue disorders) | 14 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 9
Arachnoiditis (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 3 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 5 | 5
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 23 | 23
Dysgeusia (Nervous system disorders) | 4 | 3
Dysphasia (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 2 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 47 | 31
Intracranial hemorrhage (Nervous system disorders) | 2 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 3 | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 20 | 13
Neuralgia (Nervous system disorders) | 2 | 0
Nystagmus (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 12 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 41 | 24
Seizure (Nervous system disorders) | 6 | 0
Sinus pain (Nervous system disorders) | 6 | 1
Syncope (Nervous system disorders) | 1 | 3
Tremor (Nervous system disorders) | 1 | 5
Trigeminal nerve disorder (Nervous system disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 6 | 3
Anxiety (Psychiatric disorders) | 20 | 16
Confusion (Psychiatric disorders) | 12 | 2
Depression (Psychiatric disorders) | 18 | 9
Insomnia (Psychiatric disorders) | 31 | 19
Libido decreased (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 1
Psychosis (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 4 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 10 | 5
Urinary frequency (Renal and urinary disorders) | 5 | 6
Urinary incontinence (Renal and urinary disorders) | 3 | 1
Urinary retention (Renal and urinary disorders) | 7 | 3
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 3 | 3
Urine discoloration (Renal and urinary disorders) | 1 | 2
Breast pain (Reproductive system and breast disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
Irregular menstruation (Reproductive system and breast disorders) | 4 | 3
Pelvic pain (Reproductive system and breast disorders) | 1 | 4
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 2
Scrotal pain (Reproductive system and breast disorders) | 0 | 2
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Uterine pain (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 | 2
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 20
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 19 | 14
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 7
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 3
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 11 | 9
Nail loss (Skin and subcutaneous tissue disorders) | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 12
Purpura (Skin and subcutaneous tissue disorders) | 13 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 26 | 18
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 22 | 15
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3
Flushing (Vascular disorders) | 7 | 5
Hematoma (Vascular disorders) | 5 | 2
Hot flashes (Vascular disorders) | 1 | 4
Hypertension (Vascular disorders) | 7 | 2
Hypotension (Vascular disorders) | 13 | 6
Phlebitis (Vascular disorders) | 2 | 1
Thromboembolic event (Vascular disorders) | 23 | 10
Vascular disorders - Other, specify (Vascular disorders) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes